CLINICAL TRIAL: NCT02107105
Title: Prospective Evaluation of Quality of Life and Utilities Following Surgical Treatment of Rectal Cancer
Brief Title: Evaluation of Quality of Life and Utilities Following Surgical Treatment of Stage I-IV Rectal Cancer
Status: Suspended | Type: Observational
Why Stopped: PI requested
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0631; NCI-2020-07835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0631 (Other: M D Anderson Cancer Center); K07CA133187 (NIH)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Rectal Adenocarcinoma; Stage I Rectal Cancer AJCC v8; Stage II Rectal Cancer AJCC v8; Stage IIA Rectal Cancer AJCC v8; Stage IIB Rectal Cancer AJCC v8; Stage IIC Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete quality of life questionnaires over 20-30 minutes at baseline, 6 and 12 months after surgery, and 2, 3, 4, and 5 years after surgery.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete quality of life questionnaire
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete quality of life questionnaire

SUMMARY:
This study evaluates quality of life and utilities following surgical treatment of stage I-IV rectal cancer. This study may help researches learn more about quality of life in patients who have or have had rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess post-treatment related health state utilities among patients with rectal cancer after treatment at 2 years.

SECONDARY OBJECTIVES:

I. To longitudinally compare the effects of treatment on quality of life and utilities among patients treated with or without (neo)adjuvant radiation therapy.

II. To characterize the impact of treatment on quality of life and utilities among patients with rectal cancer.

III. To assess changes in quality of life and utilities among patients treated for rectal cancer over time.

OUTLINE:

Patients complete quality of life questionnaires over 20-30 minutes at baseline, 6 and 12 months after surgery, and 2, 3, 4, and 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically proven adenocarcinoma of the rectum (stage I - IV) that is planned to be treated by surgical resection performed with curative intent, or who has already received surgical treatment
* Patient must sign an approved informed consent document and have the literary and physical ability to complete the questionnaire in English

Exclusion Criteria:

* Patient has been treated with pelvic radiation therapy for a diagnosis other than rectal cancer
* Patient has a concurrent cancer diagnosis at the time of consent
* Patient has recurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with stave I-IV rectal adenocarcinoma at the Colorectal Clinic at M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2014-05-16 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Health state utilities | At 24 months post-surgery
  A health state utility is the degree of preference that individuals or society has for a particular health state or condition.

CONTACTS AND LOCATIONS:
Overall Officials: George J Chang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org